CLINICAL TRIAL: NCT03415282
Title: Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of RVT-501 Topical Ointment in Pediatric Patients With Atopic Dermatitis
Brief Title: Open-Label Study of RVT-501 Topical Ointment in Pediatric Patients With Atopic Dermatitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dermavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Organization: Dermavant Sciences, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-501-2007
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — methyl 4-(((3-(6,7-dimethoxy-2-(methylamino)quinazolin-4-yl)phenyl)amino)carbonyl)benzoate; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label treatment arm (Experimental): Open-label treatment arm - patients will receive RVT-501 0.5% twice daily (BID) for 4 weeks.
  Interventions: Drug: RVT-501 0.5% topical ointment

INTERVENTIONS:
Drug: RVT-501 0.5% topical ointment — RVT-501 0.5% topical ointment twice daily (BID) for 4 weeks.

SUMMARY:
This is a multicenter, open-label Phase 1b study in pediatric patients age 2-11 years old with extensive atopic dermatitis.

DETAILED DESCRIPTION:
The purpose of this multicenter, open-label study is to evaluate the safety, tolerability, and pharmacokinetics of RVT-501 0.5% topical ointment administered twice daily (BID) for 4 weeks in pediatric patients age 2-11 years of age with extensive atopic dermatitis. The efficacy of RVT-501 will also be evaluated as a secondary objective in these patients. The study will consist of three phases: Screening (up to 30 days), Treatment Phase (28 days), and Follow-up (7-10 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female pediatric patients aged 2 to 11 with confirmed diagnosis of atopic dermatitis by Hanifin and Rajka criteria.
2. Patients with atopic dermatitis covering > 25% of the body surface area and with an Investigator Global Assessment of disease severity of 2 or greater at baseline.
3. Minimum body weight of 10 kg.
4. Females of childbearing potential and male patients, who are engaging in sexual activity that could lead to pregnancy, must use the following adequate birth control methods while on study and for 2 weeks after stopping study drug. Acceptable contraception methods are:

   * Male or male partner with vasectomy OR
   * Male condom, AND partner use of one of the contraceptive options below:

     * Spermicide
     * Contraceptive subdermal implant that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label
     * Intrauterine device or intrauterine system that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label
     * Oral Contraceptive, either combined or progestogen alone
     * Injectable progestogen
     * Contraceptive vaginal ring
     * Percutaneous contraceptive patches

   These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The Investigator is responsible for ensuring that patients understand how to properly use these methods of contraception.

   Nonchildbearing potential is defined as premenarchal or premenopausal females with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy; or hysteroscopic sterilization. Documented verbal history from the patient is acceptable.

   Patients who are abstinent are eligible, but they must use one of the birth control methods listed above if they start engaging in sexual activity that could lead to pregnancy during the study.

   Female patients of childbearing potential must have a negative pregnancy test at screening and Baseline (Day 0).
5. History of atopic dermatitis and stable disease for at least 1 month according to the patient or caregiver.
6. Patient or patient's parent(s)/legal representative must be capable of giving written informed consent or verbal assent, as applicable, which includes compliance with the requirements and restrictions listed in the consent/assent form; written informed consent must be obtained prior to any study related procedures.

Exclusion Criteria:

1. A positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody result, or positive human immunodeficiency virus (HIV) antibody at Screening.
2. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5x the upper limit of normal (ULN).
3. Screening total bilirubin > 1.5x ULN; total bilirubin > ULN and ≤ 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
4. Patients with a skin condition such as Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo, psoriasis, severe acne, connective tissue disorder, or Netherton's syndrome, or any other disease that could impact study evaluations.
5. Use of any prohibited medication. Prohibited concomitant medications, therapy, etc. during the defined period are as listed in the bullets below. If a patient requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the Investigator and medical monitor.

   * From 6 months prior to the first application of study drugs to the completion of the Follow-up visit or discontinuation:

     * Biological products that might have significantly affected the evaluation of atopic dermatitis condition (e.g., tumor necrosis factor [TNF] inhibitors, anti-immunoglobulin [Ig]E antibodies, anti-CD20 antibodies, anti-interleukin [IL]-4 receptor).
   * From 28 days prior to the first application of study drug until the completion of the Follow-up visit or discontinuation:

     * Corticosteroid preparations (oral, injection, and suppository preparations) and topical corticosteroids that were classified as super-high potency (clobetasol propionate). Eye drops and nasal preparations are allowed. Inhaled preparations are allowed if used for a stable condition and at stable dose for ≥ 28 days before Screening, and are continued at the same dose throughout the study.
     * Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, etc.);
     * Excessive sun exposure, tanning booth, other ultraviolet (UV) light source and phototherapy including psoralen and ultraviolet A (PUVA) therapy.
   * From 14 days prior to the first application of the study drug to the completion of the

   Follow-up visit or discontinuation:
   * Herbal medicines for atopic dermatitis (topical and oral preparations), unless specifically approved by the Sponsor;
   * Eucrisa™ (crisaborole) and any other topical phosphodiesterase 4 (PDE4) inhibitor;
   * Tacrolimus and pimecrolimus cream and/or ointment;
   * Topical corticosteroids that were classified as low, medium, or high potency (e.g., fluocinonide, triamcinolone acetonide, desonide, hydrocortisone). Eye drops and nasal preparations are allowed.

     * From 7 days prior to the first application of the study drug to the completion of the Follow- up visit or discontinuation:
   * Oral or intravenous antibiotics, antifungal or antivirus medications
   * Antihistamines/anti-allergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine).

   NOTE: The following antihistamines are allowed:
   * Loratadine, fexofenadine hydrochloride, cetirizine hydrochloride
6. Pregnant or lactating females.
7. History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or medical monitor, contraindicates their participation.
8. The patient has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
9. Current or a history of cancer within 5 years.
10. Patients with active infection in atopic dermatitis areas requiring antibiotics, antifungals, or antiviral agents within 7 days of Baseline (Day 0).
11. Patients with pruritus due to conditions other than atopic dermatitis that, in the opinion of the Investigator, would either interfere with study evaluations or affect the safety of the patient.
12. Patients with advanced disease or recent abnormal laboratory test values that could affect the safety of the patient or the implementation of this study.
13. History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to PDE4 inhibitors.
14. Prior exposure to RVT-501.
15. Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities or laboratory abnormalities that will affect the health of the patient or interfere with interpretation of the results.
16. The patient has excessive sun exposure, is planning a trip to a sunny climate that would involve excessive sun exposure, or used tanning booths within 28 days prior to Baseline (Day 0) or is not willing to minimize natural and artificial sunlight exposure during the study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-07-24 (Estimated); Study Completion 2018-08-07 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (local and systemic) | 28 days
  Adverse events will be coded using the most current release of MedDRA® (Medical Dictionary for Regulatory Activities). The number and proportion of subjects with adverse events will be summarized by treatment, system organ class, and preferred term for all adverse events, all adverse events considered by the investigator to be related to study drug, all serious adverse events, and all adverse events leading to study drug discontinuation
Laboratory values | 28 days
  Selected laboratory data will be summarized by the observed data and by the change from baseline (as appropriate) across time. Incidence of treatment emergent laboratory values that are considered clinically significantly abnormal will be summarized by treatment group.
Vital signs | 28 days
  Vital signs will be measured in supine or semi-supine position after a 5 minute rest and will include systolic and diastolic blood pressure and pulse rate. Vital sign data will be listed by subject and summarized by treatment.
Plasma concentrations of RVT-501 | 28 days
  PK samples will be collected at week 1 pre-dose, 2-4 hours post-dose, and 6-8 hours post dose for all subjects. At week PK samples will be collected pre-dose. RVT-501 will be measured in plasma by validated assay in all subjects to confirm exposure. These plasma concentrations will be listed by metabolite, subject, treatment, and time; and will be summarized by analyte and time. If data permit, RVT-501 and M11 concentrations will be summarized descriptively at each collection time point.
Plasma concentrations of M11 metabolite | 28 days
  PK samples will be collected at week 1 pre-dose, 2-4 hours post-dose, and 6-8 hours post dose for all subjects. At week 4 PK samples will be collected pre-dose. The M11 metabolite will be measured in plasma by validated assay in all subjects to confirm exposure. These plasma concentrations will be listed by metabolite, subject, treatment, and time; and will be summarized by metabolite, treatment and time. If data permit, RVT-501 and M11 concentrations will be summarized descriptively at each collection time point.

SECONDARY OUTCOMES:
Efficacy - Investigators Global Assessment (IGA) | 28 days
  Efficacy will be evaluated as the change from Baseline in IGA score.
Efficacy - 2-point improvement in IGA | 28 days
  Efficacy will be evaluated by the proportion of patients who achieve an IGA of 0 or 1 with at least a 2-point improvement from Basline
Efficacy - IGA of 0 or 1 at study end | 28 days
  Efficacy will be evaluated by the proportion of patients who achieve an IGA of 0 or 1 at Week 4.
Efficacy - Eczema Area and Severity Index (EASI) score | 28 days
  Efficacy will be evaluated as the change from Baseline in EASI score.
Efficacy - EASI-50 | 28 days
  Efficacy will be evaluated by the proportion of patients who achieve at least a 50% reduction from Baseline EASI (EASI-50) at Week 4.
Efficacy - Peak Pruritus Numeric Rating Scale (NRS) | 28 days
  Efficacy will be evaluated as the change from Baseline in Peak Pruritus as measured with the NRS at Week 4.
Efficacy - Body Surface Area (BSA) | 28 days
  Efficacy will be evaluated as the change from Baseline in BSA affected by disease at Week 4.
Efficacy - Patient/caregiver reported itch severity (local) | 28 days
  The patient or their caregiver will assess itch severity at the application site and efficacy will be determined as a change from Baseline.
Efficacy - Patient/caregiver reported itch severity (global) | 28 days
  The patient or their caregiver will assess global itch severity and efficacy will be determined as change from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: James Lee, MD, PhD, Study Chair — Dermavant Sciences, Inc.
Locations (10):
- United States (10):
  - Dermavant Investigational Site, Anniston, Alabama
  - Dermavant Investigational Site, Irvine, California
  - Dermavant Investigational Site, Jacksonville, Florida
  - Dermavant Investigational Site, Miami, Florida
  - Dermavant Investigational Site, Stockbridge, Georgia
  - Dermavant Investigational Site, Indianapolis, Indiana
  - Dermavant Investigational Site, Raleigh, North Carolina
  - Dermavant Investigational Site, Arlington, Texas
  - Dermavant Investigational Site, San Antonio, Texas
  - Dermavant Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official Website for Dermavant Sciences — http://dermavant.com